CLINICAL TRIAL: NCT05161910
Title: Urinary Biomarker Neutrophil Gelatinase Associated Lipocalcin (NGAL) in Early Prediction of AKI in Cirrhosis of Liver
Brief Title: ROLE OF URINARY BIOMARKER NEUTROPHIL GELATINASE ASSOCIATED LIPOCALCIN (NGAL) IN EARLY PREDICTION OF AKI IN CIRRHOSIS OF LIVER
Acronym: NGAL
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Clinical Professor, Asian Institute of Gastroenterology, India
Other Study IDs: CLD
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarkers — Kidney biomarkers appear to be useful in differential diagnosis between acute tubular necrosis (ATN) and other types of acute kidney injury (AKI) in cirrhosis, particularly hepatorenal syndrome (HRS-AKI).

SUMMARY:
Kidney dysfunction is a complex and common event in patients with liver cirrhosis. Although novel treatments have shown some promising results , acute kidney injury remains a major complication of decompensated liver cirrhosis with high morbidity and mortality rates . AKI occurs in up to 19-20% of hospitalized patients with liver cirrhosis and among the most frequent causes are prerenal azotemia (PRA), hepatorenal syndrome and acute tubular necrosis , with prevalence rates estimated around 68%, 25%, and 33%, respectively.

The introduction and widespread use of diagnostic criteria of AKI in the area of cirrhosis has contributed to an increased awareness and earlier detection of AKI. However, some important problems remain. One of the main issues is the differential diagnosis of AKI, particularly between acute tubular necrosis (ATN) and hepatorenal syndrome (HRS-AKI). This is important because treatment is different; renal replacement therapy (RRT) is used for the former, and vasoconstrictors and albumin are used for the latter.

DETAILED DESCRIPTION:
Aim of the study:

To determine utility of NGAL in chronic liver disease patients with acute kidney injury.

Objective:

1. To compare urine NGAL values in HRS and Non-HRS group.
2. To determine optimal cutoff of urine NGAL for early determination of HRS.

Plan of investigation:

All the following investigations will be done at admission for the patients who satisfy the inclusion criteria

Routine blood investigations :

CBP, LFT, PT- INR, RFT urine sodium on day 1 urine spot urine protein creatinine ratio CUE Urine c/s Urine NGAL Serum creatinine will be repeated on Day 3.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosis by combination of clinical, laboratorial, endoscopic and imaging
* Age over 18 years old
* Acute kidney injury (defined by ICA-AKI criteria)
* Agreement to participate in the study

Exclusion Criteria:

* Shock/CCF
* Age less than 18yrs •
* Underwent renal replacement therapy within the last 6 week prior to evaluation
* Prior kidney or liver transplantation
* Confirmed pregnancy
* Established CKD
* Congestive cardiac failure
* Patients who have taken diuretics in the last 48 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
To compare urine Neutrophil Gelatinase Associated lipocalcin values in Hepato renal syndrome and Non-Hepato renal syndrome group. | 12 months
  Kidney biomarkers appear to be useful in differential diagnosis between acute tubular necrosis (ATN) and other types of acute kidney injury (AKI) in cirrhosis, particularly hepatorenal syndrome (HRS-AKI)

SECONDARY OUTCOMES:
. To determine optimal cutoff of urine NGAL for early determination of HRS. | 12 months
  increase in the serum creatinine ≥ 0.3 mg/dl within 48 h or ≥ 50% from baseline value according to ICA(international club ascites) consensus document and /or urinary output ≤ 0.5 ml/kg B.W. ≥6h

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MBBS MD, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No